CLINICAL TRIAL: NCT01335698
Title: A Prospective Single Arm, Open-label, International, Multicenter Study to Evaluate the Safety, Efficacy and Pharmacokinetics of Atazanavir (ATV) Powder Boosted With Ritonavir (RTV) With an Optimized NRTI Background Therapy, in Human Immunodeficiency Virus (HIV) Infected, Antiretroviral, Naive and Experienced Pediatric Subjects From 3 Months to Less Than 11 Years.(Pediatric Atazanavir International Clinical Evaluation: the PRINCE II Study)
Brief Title: Phase IIIB Study Evaluating the Effects of Atazanavir Powder With Ritonavir in HIV-infected Pediatric Patients
Acronym: PRINCE2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI424-451; 2010-024537-23 (EudraCT Number)
Record Dates: First submitted 2011-04-13; First posted 2011-04-14 (Estimated); Results first posted 2016-02-08 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: HIV
Keywords: Pediatric
MeSH Terms: interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Stage 1: Atazanavir + Ritonavir (Experimental): Participants received atazanavir powder orally (dosed by weight: 5 to <10 kg=150 mg, 5 to <10 kg=200 mg, 10 to <15 kg=200 mg, 15 to <25 kg=250 mg, 25 to <35 kg=300 mg) once daily for 24 to 48 weeks or a weight ≥35 kg. Participants also received ritonavir once daily for 24 to 48 weeks or weight ≥35 kg in the form of 80-mg/mL solution, orally (dosed by weight 5 to <25 kg=80 mg, 25 to <35 kg=100 mg); 100-mg capsule, orally (dosed by weight 25 to <35 kg=100 mg); or 100-mg tablet, orally (dosed by weight 25 to <35 kg=100 mg)
  Interventions: Drug: Atazanavir Sulphate; Drug: Ritonavir

INTERVENTIONS:
Drug: Atazanavir Sulphate
  Other Names: Reyataz; BMS-232632
Drug: Ritonavir
  Other Names: Norvir

SUMMARY:
The purpose of this study is to describe the safety, efficacy, and pharmacokinetics of a regimen of atazanavir powder boosted with ritonavir and an optimized dual nucleoside reverse transcriptase inhibitor in pediatric patients aged ≥3 months to <11 years.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Key Inclusion Criteria:

* Confirmed HIV-1 infection diagnosed by protocol criteria
* Screening HIV RNA level ≥1000 copies/mL
* ≥3 months to <11 years of age at time of first treatment
* Antiretroviral-naive or -experienced
* At screening, all participants must have genotypic sensitivity to atazanavir and at least 2 nucleoside reverse transcriptase inhibitors (NRTIs), which must be approved for pediatric use at the local country.
* Antiretroviral-experienced patients must also have documented phenotypic sensitivity at screening to atazanavir (Fold Change in susceptibility <2.2) and to at least 2 NRTIs that are approved in their country

Key Exclusion Criteria:

* Experienced participants who received atazanavir or atazanavir/ritonavir at any time prior to study enrollment or who have a history of 2 or more protease inhibitor failures
* Antiretroviral-naïve or -experienced HIV-1-infected patients with contraindication to study medications
* Cardiac rhythm abnormalities
* Need for tenofovir
* Weight <5 or ≥35kg
* >Grade 2 abnormality in aspartate transaminase/alanine transaminase levels
* Coinfection with either hepatitis B or C virus
* Any active Centers for Disease Control and Prevention Category C clinical condition

Ages: 3 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2011-05-27 (Actual); Primary Completion 2014-09-10 (Actual); Study Completion 2018-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (27):
- United States (2):
  - Children'S National Medical Center, Washington D.C., District of Columbia
  - SUNY Upstate Medical University, Syracuse, New York
- Argentina (2):
  - Local Institution, Buenos Aires, Bs As, Buenos Aires
  - Local Institution, Bunos Aires, Buenos Aires
- Brazil (3):
  - Local Institution, Recife, Pernambuco
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Ribeirão Preto, São Paulo
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Mexico (5):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Mérida, Yucatán
  - Local Institution, Oaxaca City
  - Local Institution, Puebla City
- Local Institution, Warsaw, Poland
- Local Institution, Bucharest, Romania
- Russia (2):
  - Local Institution, Saint Petersburg
  - Local Institution, Smolensk
- South Africa (7):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Benoni, Gauteng
  - Local Institution, Coronationville, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Soweto, Gauteng
  - Local Institution, Parrow Valley, Western Cape
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Madrid
- Local Institution, Birmingham, WEST Midlands, United Kingdom

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 160 participants enrolled, 99 received treatment.
Groups:
- Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg); Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg): Stage 1: HIV-infected pediatric patients weighing 5 to <10 kg at baseline received atazanir powder formulation, 150 mg, with ritonavir oral solution, 80 mg, for 24 to 48 weeks. Patients entering Stage 2 continued Stage 1 treatment but those aged 12 years or older or weighing at least 35 kg transitioned to capsules. Treatment continued until the patient reached 18 years of age or pediatric indication is locally approved and patient meets requirements to receive appropriate formulation.
- Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg): Stage 1: HIV-infected pediatric patients weighing 10 to <15 kg at baseline received atazanir powder formulation, 200 mg, with ritozinavir oral solution, 80 mg, for 24 to 48 weeks. Patients entering Stage 2 continued Stage 1 treatment but those aged 12 years or older or weighing at least 35 kg transitioned to capsules. Treatment continued until the patient reached 18 years of age or pediatric indication is locally approved and patient meets requirements to receive appropriate formulation.
- Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg): Stage 1: HIV-infected pediatric patients weighing 15 to <25 kg at baseline received atazanir powder formulation, 250 mg, with ritozinavir oral solution, 80 mg, for 24 to 48 weeks. Patients entering Stage 2 continued Stage 1 treatment but those aged 12 years or older or weighing at least 35 kg transitioned to capsules. Treatment continued until the patient reached 18 years of age or pediatric indication is locally approved and patient meets requirements to receive appropriate formulation.
- Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg): Stage 1: HIV-infected pediatric patients weighing 10 to <15 kg at baseline received atazanir powder formulation, 300 mg, with ritozinavir capsule/tablets, 100 mg, for 24 to 48 weeks. Patients entering Stage 2 continued Stage 1 treatment but those aged 12 years or older or weighing at least 35 kg transitioned to capsules. Treatment continued until the patient reached 18 years of age or pediatric indication is locally approved and patient meets requirements to receive appropriate formulation.
Period: Treatment Stage 1
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Started | 23 | 12 | 21 | 35 | 8
Completed | 15 | 4 | 16 | 26 | 6
Not Completed | 8 | 8 | 5 | 9 | 2
Not completed — Lack of Efficacy | 3 | 1 | 3 | 3 | 1
Not completed — Adverse Event | 1 | 2 | 2 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Poor compliance/noncompliance | 0 | 1 | 0 | 2 | 0
Not completed — No longer meets study criteria | 1 | 1 | 0 | 1 | 0
Not completed — Other | 1 | 0 | 0 | 1 | 0
Period: Treatment Stage 2
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Started | 15 | 4 | 16 | 26 | 6
Completed | 4 | 1 | 11 | 18 | 5
Not Completed | 11 | 3 | 5 | 8 | 1
Not completed — Lack of Efficacy | 2 | 1 | 3 | 1 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 0 | 0
Not completed — Poor compliance/noncompliance | 1 | 0 | 1 | 3 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Capsules received at state hospital | 1 | 0 | 0 | 0 | 0
Not completed — Subject no longer meets study criteria | 0 | 0 | 0 | 1 | 0
Not completed — Switched to another formulation | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg) | Total
Number analyzed (Participants) | 23 | 12 | 21 | 35 | 8 | 99
Age, Continuous [Mean (Standard Deviation); unit: Months] | 8.4 (6.42) | 10.5 (9.21) | 37.4 (12.44) | 67.2 (16.70) | 93.4 (15.53) | 42.5 (31.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 12 | 18 | 3 | 51
  Male | 11 | 6 | 9 | 17 | 5 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 1 | 0 | 4
  Not Hispanic or Latino | 1 | 1 | 1 | 1 | 0 | 4
  Unknown or Not Reported | 22 | 10 | 18 | 33 | 8 | 91
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 2 | 12 | 13 | 3 | 32
  Black/African American | 19 | 6 | 7 | 20 | 5 | 57
  Other | 2 | 4 | 2 | 2 | 0 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 2 | 1 | 9 | 4 | 2 | 18
  South America | 1 | 1 | 1 | 4 | 1 | 8
  Africa | 20 | 10 | 8 | 21 | 5 | 64
  Europe | 0 | 0 | 3 | 6 | 0 | 9
Country [Count of Participants; unit: Participants]
  Argentina | 0 | 1 | 1 | 2 | 0 | 4
  Brazil | 0 | 0 | 0 | 1 | 0 | 1
  Chile | 1 | 0 | 0 | 1 | 1 | 3
  Mexico | 1 | 1 | 7 | 4 | 2 | 15
  Poland | 0 | 0 | 1 | 0 | 0 | 1
  Romania | 0 | 0 | 0 | 1 | 0 | 1
  Russia | 0 | 0 | 1 | 3 | 0 | 4
  South Africa | 20 | 10 | 8 | 21 | 5 | 64
  Spain | 0 | 0 | 1 | 2 | 0 | 3
  United States | 1 | 0 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died and With Adverse Events (AEs) Leading to Discontinuation, Hyperbilirubinemia, Jaundice, First-degree Arterioventricular Block, Tachycardia, and Rash on ATV Powder
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment.
Time Frame: Day one to week 300 (approximately 22-Jan-2018)
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 23 | 12 | 21 | 35 | 8
Participants
  Deaths | 0 | 0 | 0 | 0 | 0
  AEs leading to discontinuation | 3 | 2 | 2 | 2 | 1
  Hyperbilirubinemia related adverse events | 2 | 0 | 9 | 7 | 0
  Jaundice | 0 | 0 | 3 | 3 | 0
  Atrioventricular block, first degree | 0 | 0 | 0 | 1 | 0
  Tachycardia | 0 | 0 | 1 | 0 | 0
  Rash | 3 | 0 | 4 | 5 | 1

2. Primary Outcome: Number of Participants Who Experienced a SAE on ATV Powder
Description: SAE= any of the the following: is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event (defined as a medical event(s) that may not be immediately life threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the subject or may require intervention [eg, medical, surgical] to prevent one of the other serious outcomes listed in the definition above.) Examples of such events include, but are not limited to, intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization
Time Frame: Day one to week 300 (approximately 22-Jan-2018)
Measure: Number; unit: participants
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 23 | 12 | 21 | 35 | 8
participants | 6 | 3 | 8 | 8 | 0

3. Primary Outcome: Number of Participants With A Center of Disease Control and Prevention (CDC) Class C AIDS Event on ATV Powder
Description: The CDC disease staging system assesses the severity of HIV disease by CD4 cell counts and by the presence of specific HIV-related conditions. CD4 counts are classified as 1: ≥500 cells/µL, 2: 200-499 cells/µL, and 3: <200 cells/µL. Children with HIV infection are also classified in each of several categories. Category N: Not symptomatic. Category A: Mildly symptomatic. Category B: Moderately symptomatic. Category C: Severely symptomatic.
Time Frame: Day one to week 300 (approximately 22-Jan-2018)
Population: All participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 23 | 12 | 21 | 35 | 8
Participants
  Pulmonary tuberculosis | 2 | 0 | 1 | 0 | 0
  Lymph node tuberculosis | 0 | 0 | 0 | 1 | 0
  Tuberculosis | 0 | 0 | 0 | 1 | 0
  Oropharyngeal Candidiasis | 1 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Grade 3-4 Abnormality on ATV Powder
Description: Criteria of the Division of AIDS for grading the severity of adult and pediatric adverse events as follows: Grade (Gr) 1=mild; Gr 2=moderate; Gr 3=severe; Gr 4=potentially life-threatening. Neutrophils (absolute) (adult and infants >7 days): Gr 1=1.000-1300/mm^3; Gr 2=750-999 mm^3; Gr 3=500-749 mm^3; Gr 4= <500 mm^3. Alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase: Gr 1=1.25-2.5*upper limit of normal (ULN); Gr 2=2.6-5.0*ULN; Gr 3=5.1-10.0*ULN; Gr 4= >10.0*ULN. Bilirubin, total (adults and infants >14 days): Gr 1=1.1-1.5*ULN; Gr 2=1.6-2.5*ULN; Gr 3=2.6-5.0*ULN; Gr 4= >5.0*ULN. Lipase: Gr 1=1.1-1.5*ULN; Gr 2=1.6-3.0*ULN; Gr 3=3.1-5.0*ULN; Gr 4= >5.0*ULN. Bicarbonate, serum low: Gr 1=16.0 mEq/L-<lower limit of normal; Gr 2=11.0-15.9 mEq/L; Gr 3=8.0-10.9 mEq/L; Gr 4= <8 mEq/L. By criteria of the World Health Organization: Amylase: Gr 1=1.0-1.39*ULN; Gr 2=1.40-2.09*ULN; Gr 3.=2.10-5.0*ULN; Gr 4= >5.0*ULN.
Time Frame: Day one to week 300 (approximately 22-Jan-2018)
Population: All participants who received at least 1 dose of study drug. n=number of participants evaluable
Measure: Number; unit: Participants
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 23 | 12 | 21 | 35 | 8
Participants
  Neutrophils (absolute): number analyzed (Participants) | 23 | 11 | 21 | 34 | 8
  Neutrophils (absolute) | 0 | 0 | 4 | 6 | 0
  Alanine aminotransferase: number analyzed (Participants) | 23 | 12 | 21 | 34 | 8
  Alanine aminotransferase | 4 | 1 | 1 | 2 | 0
  Aspartate aminotransferase: number analyzed (Participants) | 17 | 12 | 21 | 34 | 8
  Aspartate aminotransferase | 2 | 0 | 1 | 0 | 0
  Alkaline phosphatase: number analyzed (Participants) | 23 | 12 | 21 | 34 | 8
  Alkaline phosphatase | 1 | 2 | 1 | 0 | 0
  Total bilirubin: number analyzed (Participants) | 23 | 12 | 21 | 34 | 8
  Total bilirubin | 4 | 1 | 10 | 5 | 2
  Amylase: number analyzed (Participants) | 23 | 12 | 21 | 34 | 8
  Amylase | 15 | 7 | 6 | 6 | 1
  Lipase: number analyzed (Participants) | 23 | 12 | 21 | 34 | 8
  Lipase | 3 | 2 | 0 | 2 | 1
  Bicarbonate: number analyzed (Participants) | 23 | 12 | 21 | 34 | 8
  Bicarbonate | 2 | 0 | 0 | 0 | 0
  Albumin: number analyzed (Participants) | 23 | 12 | 21 | 34 | 8
  Albumin | 1 | 1 | 0 | 1 | 0
  Calcium, High: number analyzed (Participants) | 23 | 12 | 21 | 34 | 8
  Calcium, High | 0 | 0 | 0 | 1 | 0
  Chloride, Low: number analyzed (Participants) | 23 | 12 | 21 | 34 | 8
  Chloride, Low | 0 | 0 | 0 | 1 | 0
  Total Cholesterol, Fasting: number analyzed (Participants) | 11 | 7 | 15 | 26 | 6
  Total Cholesterol, Fasting | 0 | 0 | 1 | 0 | 0
  LDL Cholesterol, Fasting: number analyzed (Participants) | 10 | 3 | 15 | 26 | 6
  LDL Cholesterol, Fasting | 0 | 0 | 1 | 0 | 0
  Glucose, Fasting, Low: number analyzed (Participants) | 14 | 7 | 17 | 28 | 8
  Glucose, Fasting, Low | 0 | 0 | 1 | 0 | 0

5. Secondary Outcome: Number of Participants With HIV RNA <50 Copies/mL and <400 Copies/mL in the Week 24 Atazanavir Powder Cohort and the Eligible Week 48 Atazanavir Powder Cohort
Description: Virologic success includes patients with HIV RNA <50 copies/mL. Two cohorts were assessed: The Atazanavir Powder Cohort=patients who received treatment and did not switch to capsule before analysis Week 24 or before their HIV RNA Week 24 assessment, and the Eligible Week 48 Atazanavir Powder Cohort=patients who initiated study treatment at least 48 weeks before last person last visit and did not switch to capsule before analysis Week 48 or before their HIV RNA Week 48 assessment.
Time Frame: Day 1 of treatment to weeks 24 and 48
Population: For efficacy of atazanavir powder to Week 24: Atazanavir Powder Cohort. For efficacy of atazanavir powder efficacy to Week 48 (n): Eligible Week 48 Atazanavir Powder Cohort
Measure: Number; unit: Participants
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 23 | 12 | 21 | 35 | 8
Participants
  Week 24: HIV RNA<50 copies/mL | 10 | 2 | 10 | 19 | 5
  Week 24: HIV RNA<400 copies/mL | 15 | 5 | 15 | 24 | 6
  Week 48: HIV RNA<50 copies/mL | 11 | 0 | 6 | 18 | 1
  Week 48:HIV RNA<400 copies/mL | 14 | 1 | 14 | 22 | 1

6. Secondary Outcome: Mean Change From Baseline in HIV RNA on ATV Powder
Description: Human immunodeficiency virus ribonucleic acid (HIV RNA) change from baseline using observed values
Time Frame: Baseline to Weeks 24 and 48
Population: All participants who received at least 1 dose of study drug. n=participants with both baseline and time point results
Measure: Mean (Standard Error); unit: Log copies per millileter
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 23 | 12 | 21 | 35 | 8
Log copies per millileter
  Week 24 | -2.10 (0.2863) | -3.07 (0.4780) | -2.69 (0.2257) | -2.66 (0.1550) | -2.24 (0.3821)
  Week 48: number analyzed (Participants) | 23 | 12 | 21 | 35 | 1
  Week 48 | -2.31 (0.3174) | -4.06 (0.1649) | -2.91 (0.1883) | -2.70 (0.1269) | -3.97 (NA) — Only 1 participant in this arm was eligible for evaluation at this time point

7. Secondary Outcome: Mean Change From Baseline in CD4 Percent on ATV Powder
Description: Change in CD4 percent using observed values
Time Frame: Baseline to Weeks 24 and 48
Population: All participants with both baseline and time point results; n=number of participants evaluable at time point
Measure: Mean (Standard Error); unit: Percent Change
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 23 | 12 | 21 | 35 | 8
Percent Change
  Week 24: number analyzed (Participants) | 17 | 4 | 12 | 23 | 6
  Week 24 | 5.1 (1.521) | 4.0 (1.581) | 5.4 (2.448) | 6.3 (1.280) | -0.3 (4.349)
  Week 48: number analyzed (Participants) | 12 | 0 | 9 | 19 | 1
  Week 48 | 2.8 (3.167) |  | 8.9 (2.182) | 7.5 (1.825) | 1.0 (NA) — Only one participant was analyzed

8. Secondary Outcome: CD4 Cell Count Changes From Baseline on ATV Powder
Description: CD4 cell count change from baseline using observed values
Time Frame: Baseline to Weeks 24 and 48
Population: All participants with both baseline and time point results
Measure: Mean (Standard Error); unit: Cells/mm^3
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 10 | 1 | 13 | 27 | 8
Cells/mm^3
  Week 24 | 218.7 (259.102) | 67.8 (425.659) | 247.1 (110.739) | 246.1 (72.044) | 145.8 (78.443)
  Week 48: number analyzed (Participants) | 10 | 0 | 13 | 27 | 1
  Week 48 | -409.8 (437.686) |  | 400.0 (156.021) | 335.4 (108.925) | 213.0 (NA) — Only one participant was analyzed

9. Secondary Outcome: Number of Participants With Emergent Genotypic Substitutions on ATV Powder Through Week 48
Description: Newly emergent substitutions are on-treatment substitutions that were not detected at baseline.Viral rebound in the resistance analysis was defined as: Less than a 1 log10 drop from baseline in plasma HIV RNA level by Week 16, confirmed by a second plasma HIV RNA level redrawn within 2 and 4 weeks from original sample. Or, a plasma HIV RNA level >200 c/mL after Week 24, confirmed by a second plasma HIV RNA level redrawn within 2 and 4 weeks from original sample. Or, repeated plasma HIV RNA level ≥50 c/mL after Week 48. Viral rebound was defined as a plasma HIV RNA level ≥400 c/mL at any time in a patient who had previously achieved a plasma HIV RNA level <50 c/mL. Or, a plasma HIV RNA level ≥50 c/mL and <1,000 c/mL followed by a return to virologic suppression was considered a viral blip and not a viral rebound. NRTI=nucleoside reverse transcriptase inhibitor
Time Frame: Baseline through Week 48
Population: All participants with virologic failure.
Measure: Number; unit: Participants
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 200 mg + Ritonavir, 80 mg (Weight: 10 to <15 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 10 | 2 | 10 | 13 | 1
Participants
  Any PI substitutions | 4 | 0 | 4 | 3 | 0
  Any IAS-USA PI substitutions | 1 | 0 | 2 | 0 | 0
  Any select RT substitutions | 2 | 1 | 2 | 1 | 0
  NRTI | 1 | 1 | 2 | 1 | 0

10. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: To describe the PK profile of ATV powder formulation with RTV in pediatric subjects weighing 25 - < 35 kg and/or 6 to < 11 years of age and for the new 5 - < 10 kg cohort (200 mg ATV and 80 mg RTV) in terms of ATV Cmax
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 12 | 17 | 8
ng/mL | 5776.70 (3417.208) | 5644.12 (3093.516) | 4893.75 (2523.959)

11. Secondary Outcome: Minimum Plasma Concentration (Cmin)
Description: To describe the PK profile of ATV powder formulation with RTV in pediatric subjects weighing 25 - < 35 kg and/or 6 to < 11 years of age and for the new 5 - < 10 kg cohort (200 mg ATV and 80 mg RTV) in terms of ATV Cmin
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 12 | 17 | 8
ng/mL | 718.90 (432.747) | 857.06 (599.221) | 1030.64 (1070.932)

12. Secondary Outcome: Area Under the Concentration-Time Curve [AUC(TAU)]
Description: To describe the PK profile of ATV powder formulation with RTV in pediatric subjects weighing 25 - < 35 kg and/or 6 to < 11 years of age and for the new 5 - < 10 kg cohort (200 mg ATV and 80 mg RTV) in terms of ATV AUC
Time Frame: Baseline to Week 2
Measure: Mean (Standard Deviation); unit: ng.h./mL
Arm/Group | Atazanavir, 150 mg + Ritonavir, 80 mg (Weight: 5 to <10 kg) | Atazanavir, 250 mg + Ritonavir, 80 mg (Weight: 15 to <25 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: 25 to <35 kg)
Number analyzed (Participants) | 12 | 17 | 8
ng.h./mL | 49387.12 (26890.782) | 59671.80 (31706.655) | 56356.00 (35233.024)

ADVERSE EVENTS:
Arm/Group | B/L Weight 5 to lt 10kg (ATV 150mg) | B/L Weight 5 to lt 10kg (ATV 200mg) | B/L Weight 10 to lt 15kg | B/L Weight 15 to lt 25kg | B/L Weight 25 to lt 35kg
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/12 | 0/21 | 0/35 | 0/8
Serious Adverse Events (participants affected / at risk) | 6/23 | 3/12 | 8/21 | 10/35 | 0/8
Other Adverse Events (participants affected / at risk) | 22/23 | 10/12 | 19/21 | 31/35 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/L Weight 5 to lt 10kg (ATV 150mg) (N=23) | B/L Weight 5 to lt 10kg (ATV 200mg) (N=12) | B/L Weight 10 to lt 15kg (N=21) | B/L Weight 15 to lt 25kg (N=35) | B/L Weight 25 to lt 35kg (N=8)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Dysentery (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 1 | 0 | 0
Hepatitis a (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Infective corneal ulcer (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pertussis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0
Pneumonitis chemical (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Accidental exposure to product (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/L Weight 5 to lt 10kg (ATV 150mg) (N=23) | B/L Weight 5 to lt 10kg (ATV 200mg) (N=12) | B/L Weight 10 to lt 15kg (N=21) | B/L Weight 15 to lt 25kg (N=35) | B/L Weight 25 to lt 35kg (N=8)
Anaemia (Blood and lymphatic system disorders) | 8 | 2 | 0 | 2 | 0
Basophilia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 2 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 2 | 2 | 0
Goitre (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 0 | 2 | 1
Iritis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Myopia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Dental caries (Gastrointestinal disorders) | 4 | 1 | 3 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 0 | 3 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 7 | 1 | 6 | 9 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 3 | 0 | 8 | 4 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 6 | 2 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 3 | 3 | 0
Ocular icterus (Hepatobiliary disorders) | 1 | 0 | 2 | 1 | 0
Acarodermatitis (Infections and infestations) | 6 | 0 | 1 | 3 | 0
Body tinea (Infections and infestations) | 0 | 3 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 2 | 3 | 0
Bronchitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Candida nappy rash (Infections and infestations) | 8 | 2 | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 2 | 0 | 1 | 4 | 0
Ear infection (Infections and infestations) | 0 | 0 | 2 | 2 | 0
Fungal skin infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 14 | 3 | 11 | 8 | 2
Helminthic infection (Infections and infestations) | 7 | 2 | 0 | 1 | 0
Impetigo (Infections and infestations) | 7 | 0 | 2 | 2 | 1
Influenza (Infections and infestations) | 1 | 0 | 2 | 4 | 1
Lower respiratory tract infection (Infections and infestations) | 7 | 5 | 1 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 8 | 6 | 0
Oral candidiasis (Infections and infestations) | 9 | 4 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Otitis media (Infections and infestations) | 6 | 3 | 0 | 3 | 1
Otitis media acute (Infections and infestations) | 7 | 0 | 0 | 3 | 1
Pharyngitis (Infections and infestations) | 2 | 0 | 6 | 7 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 1 | 1 | 1
Pneumonia (Infections and infestations) | 4 | 1 | 1 | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Tinea capitis (Infections and infestations) | 7 | 1 | 3 | 4 | 0
Tonsillitis (Infections and infestations) | 3 | 1 | 1 | 3 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 16 | 5 | 5 | 10 | 2
Urinary tract infection (Infections and infestations) | 3 | 1 | 0 | 2 | 1
Varicella (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Varicella zoster virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 3 | 1 | 2 | 2 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 4 | 0 | 0 | 1 | 1
Foreign body in ear (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 2 | 0
Amylase increased (Investigations) | 2 | 1 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 1 | 0 | 0
Head lag (Investigations) | 2 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 1 | 1 | 0 | 0
Transaminases increased (Investigations) | 2 | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 1 | 2 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 3 | 2
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Product taste abnormal (Product Issues) | 0 | 0 | 0 | 0 | 1
Pica (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0 | 10 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0 | 4 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 2 | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5 | 3 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 5 | 2 | 2 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Urticaria chronic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysmorphism (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
Strabismus (Eye disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral rash (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (2):
  • Study Protocol (2014-04-15): https://cdn.clinicaltrials.gov/large-docs/98/NCT01335698/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT01335698/SAP_001.pdf